CLINICAL TRIAL: NCT01296945
Title: Nutrition Knowledge for Spanish-speaking Parents: Evaluation of Paper Handouts, Computer Modules and Web Modules
Brief Title: Nutrition Knowledge for Spanish-speaking Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Darcy Thompson, Assistant Professor of Pediatrics, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: NA_00045360
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Obesity; Dental Caries
MeSH Terms: conditions — Obesity; Dental Caries | interventions — Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Kiosk (Active Comparator)
  Interventions: Other: Kiosk
- Paper (Active Comparator)
  Interventions: Other: paper
- Kiosk PLUS paper (Active Comparator)
  Interventions: Other: Kiosk PLUS paper
- kiosk PLUS web (Active Comparator)
  Interventions: Other: Kiosk PLUS web

INTERVENTIONS:
Other: Kiosk — Touchscreen computer containing three educational modules in Spanish on infant/toddler juice intake, milk, and solid/foods
  Arms: Kiosk
Other: paper — Participants will receive a paper handout with nutrition educational information.
  Arms: Paper
Other: Kiosk PLUS paper — Individuals will use the 3 computer modules on a touchscreen and receive the information on a paper handout.
  Arms: Kiosk PLUS paper
Other: Kiosk PLUS web — Participants will utilize the 3 modules on the touchscreen computer and be given a piece of paper that includes information on how to see this information again on the internet. Participants will be asked to view the modules on the web.
  Arms: kiosk PLUS web

SUMMARY:
Providing child nutrition information is a major goal of every pediatric well-child visit. Unfortunately, due to a wide array of issues, doing this effectively during clinic visits is challenging and insufficient. It is because of this that some have looked for innovative ways to enhance the delivery of this information. One such way is the use of touch screen computer programs containing nutritional information. Several studies have documented the value of patients receiving health information in such a manner.

Nonetheless, the use of this medium has not been well studied in Spanish-speaking care providers of young children. The investigators recently conducted a study that evaluated user's perception of the usability of such technology, finding that most users thought that the touchscreen was easy to use, despite their low computer confidence levels. The investigators also evaluated the impact of using nutrition modules on user's nutrition knowledge, finding that immediately after use; participant's nutrition knowledge was improved. I now propose to evaluate this technology further through a 4 armed randomized controlled trial. The goal here is to evaluate the longer term impact of the educational modules on nutrition knowledge and the impact, if any, of additional web access to the modules, on longer term knowledge. A secondary goal is to better understand nutritional habits in this population and perceptions of weight.

ELIGIBILITY:
Inclusion Criteria:

* Self identify as Latino/a
* Spanish-speaking
* Over 18 years old
* Primary caregiver to a child 2 years old and under

Exclusion Criteria:

* Child 2 years old and under has significant medical issue requiring special nutrition needs, e.g. g-tube or feeding tube dependent, severe food allergies.
* Person has used the nutrition modules before in prior studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Knowledge score | Day 14
  Knowledge score on the nutrition survey will be compared across groups at this time point.

SECONDARY OUTCOMES:
knowledge score | Day 1
  Knowledge score on the nutrition survey will be compared between the paper group and the kiosk group.
Knowledge score | 2 months
  Knowledge score on the nutrition survey will be compared across groups at this time point - 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy A Thompaon, MD, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States